CLINICAL TRIAL: NCT06940154
Title: A Phase 2, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Rademikibart as an Add-on Treatment for Acute Exacerbation in Participants With Chronic Obstructive Pulmonary Disease and Type 2 Inflammation
Brief Title: Rademikibart Add-on Treatment of an Acute COPD Exacerbation (Seabreeze STAT COPD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-201-207
Record Dates: First submitted 2025-04-03; First posted 2025-04-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: COPD Acute Exacerbation
Keywords: COPD; chronic obstructive pulmonary disease; rademikibart; Connect Biopharma; CBP-201; COPD exacerbation; type 2 inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Rademikibart (Experimental)
  Interventions: Combination Product: Rademikibart in prefilled syringe
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo in prefilled syringe

INTERVENTIONS:
Combination Product: Rademikibart in prefilled syringe — Participants receive 600 mg (4mL) of rademikibart administered subcutaneously.
  Other Names: CBP-201
  Arms: Rademikibart
Drug: Matching placebo in prefilled syringe — Participants receive 4mL of placebo matched to rademikibart administered subcutaneously.
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter study in adult participants with an acute COPD exacerbation and type 2 inflammation

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group, interventional trial in participants with an acute COPD exacerbation with type 2 inflammation in the urgent healthcare setting to compare rademikibart plus standard therapy to standard therapy (plus placebo).

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed COPD with duration of ≥12 months.
* Must have experienced at least 1 COPD exacerbation requiring the use of systemic corticosteroids.
* Participants in a stable condition must have a documented historical peripheral blood eosinophil count of ≥250 cells/μL and/or FeNO ≥ 25 ppb.
* Current or former smoker with a history of smoking of ≥10 pack-years.
* Current acute COPD exacerbation requiring an urgent healthcare visit for treatment.
* Peripheral blood eosinophil count of ≥300 cells/μL as part of the assessment of the index acute COPD exacerbation.
* Requires systemic corticosteroids as standard of care treatment in the urgent healthcare setting for the current acute COPD exacerbation.

Exclusion Criteria:

* Regular use of immunosuppressive medication 12 weeks or 5 half-lives prior to randomization, whichever is longer.
* Current diagnosis or a history of asthma, according to the Global Initiative for Asthma; or participants with a current diagnosis or history of Asthma COPD Overlap Syndrome.
* Other respiratory disorders that might compromise the safety of the participant or affect the interpretation of the results.
* Unstable ischemic heart disease, cardiomyopathy, heart failure (New York Heart Association Class III or IV), uncontrolled hypertension. Cardiac arrhythmias including paroxysmal atrial fibrillation.
* Transient ischemic attack or stroke <6 months from Screening Visit; hospitalization for any cardiovascular or cerebrovascular event <6 months from Screening Visit.
* Known or suspected history of immunosuppression.
* History of known immunodeficiency disorder or hepatitis B or C.
* History of alcohol abuse and/or drug abuse.
* Recent history of cancer except basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success.
* Chronic treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for >15 hours a day.
* Participants on long-term macrolide.
* Current acute COPD exacerbation for which SoC was started >48 hours prior to Screening.
* A recent chest X-ray or computed tomography (CT) scan at Screening reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD, or a clinically significant pulmonary infection identified by chest X-ray (CT scan).
* Female participant who is pregnant, lactating or breast-feeding, or has a positive urinary β-hCG test prior to randomization.
* Receipt of any marketed nonbiologic drug that modulates type 2 cytokines 30 days or 5 half-lives prior to randomization, whichever is longer.
* Receipt of any marketed or any investigational biologic for COPD or other diseases within 16 weeks or 5 half-lives prior to randomization, whichever is longer.
* Live, attenuated vaccinations within 4 weeks prior to randomization or planned live, attenuated vaccinations during the trial.
* Treatment with oral corticosteroids and/or hospitalization for an exacerbation of COPD completed less than 4 weeks prior to randomization.

The above inclusion and exclusion criteria are not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate | 28 days
  Treatment failure is defined as death due to any cause, (re)admission to a hospital for COPD, ED (re)visit or unscheduled medical visit for worsening of COPD symptoms, or the necessity to intensify pharmacologic treatment (including second course of systemic steroids for COPD exacerbation) within 28 days after randomization.

SECONDARY OUTCOMES:
Rate of new moderate and severe COPD exacerbations over the 28 days after randomization | 28 days
Time to the first new moderate or severe COPD exacerbation in the 28 days after randomization | 28 days
Mean change from baseline (CFB) in EXACT-PRO score | Week 1, Week 2, and Week 4
  Mean CFB in clinical respiratory symptoms of COPD using the E-RS: COPD (Evaluating Respiratory Symptoms in COPD) comprised in the EXACT-PRO through Week 1, Week 2, and Week 4. The Exacerbations of Chronic Pulmonary Disease Tool - Patient-Reported Outcome (EXACT-PRO) is a PRO instrument designed to capture information on the occurrence, frequency, severity, and duration of exacerbations of disease in patients with COPD.
Absolute CFB in post-BD FEV1 at Day 3, Week 1, and Week 4 | Day 3, Week 1, and Week 4
  Absolute change from baseline in post-bronchodilator forced expiratory volume (FEV1) at Day 3, Week 1, and Week 4
Incidence of adverse events (AEs), including serious adverse events (SAEs), adverse event of special interest (AESIs), and drug-induced liver injury (DILI) reported | 56 days
Incidence of unanticipated adverse device effects (UADEs) | 56 days
Incidence of injection site reactions | 56 days

CONTACTS AND LOCATIONS:
Locations (36):
- United States (14):
  - University of Alabama at Birmingham Lung Health Center, Birmingham, Alabama
  - Amicis Research Center, Valencia, California
  - National Jewish Health, Denver, Colorado
  - Synergy Healthcare, Bradenton, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Pharmax Research of South Florida, Inc., Miami, Florida
  - Health Synergy Clinical Research, LLC, West Palm Beach, Florida
  - Primeway Clinical Research Group, Fayetteville, Georgia
  - Pivotal Research Solutions, Stonecrest, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Duke Asthma, Allergy, and Airway Center, Durham, North Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Inquest Clinical Research, Baytown, Texas
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
- Investigaciones en Patologias, San Miguel de Tucumán, Tucumán Province, Argentina
- Australia (5):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Institute for Respiratory Health, Nedlands, Western Australia
- Georgia (6):
  - "NCTLD National Center for Tuberculosis and Lung Disease" JSC, Tbilisi, NSW
  - LLC "Israel-Georgian Medical Research Clinic Healthycore", Tbilisi
  - Acad. Chapidze Emergency Cardiology Center LLC, Tbilisi
  - Acad. G. Chapidze Emergency Cardiology Center, Tbilisi
  - Caucasus Medical Center, Tbilisi
  - LLC Diacor, Tbilisi
- Serbia (5):
  - Clinical Hospital Center "Dragisa Misovic - Dedinje", Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
  - Institute for Pulmonary Diseases and Tuberculosis Nis, Niš
  - Health Center Uzice, Užice
- United Kingdom (5):
  - Medicines Evaluation Unit Ltd., Wythenshawe, Greater Manchester
  - Queen Elizabeth hospital Birmingham, Birmingham
  - University Hospitals Birmingham NHS Foundation Trust Birmingham Heartlands Hospital, Birmingham
  - Guy's and St Thomas NHS Foundation Trust, London
  - Salford Royal Hospital - Northern Care Alliance NHS Foundation Trust Barnes Clinical Research Facility, Salford

IPD SHARING:
Plan to Share IPD: No